CLINICAL TRIAL: NCT07268274
Title: Metabolism and the Impact of Protein Intake in Chronic Critically Ill Adult Patients: Protocol for a Unicentric Prospective Cohort Study (MetaChronic Study)
Brief Title: Metabolic Trajectories and Protein Intake in Long-Stay Ventilated Intensive Care Unit (ICU) Patients
Acronym: MetaChronic
Status: Active, not recruiting | Type: Observational
Sponsor: Universidade do Algarve (Other)
Responsible Party: Principal Investigator, Sílvia Margarida Correia de Castro, Principal Investigator, Intensive Care Physician, Universidade do Algarve
Other Study IDs: UAlg_a81228_SCastro
Record Dates: First submitted 2025-11-15; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Adult ICU Patients
Keywords: Metabolism; Chronic critically ill adult patients; Nutrition; inflammation
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Long-Stay critically ill patients: This cohort includes critically ill adults who remain in the Intensive Care Unit (ICU) for more than 7 days and receive invasive mechanical ventilation for at least 48 hours. Patients are monitored according to routine clinical practice. Resting energy expenditure is assessed by serial indirect calorimetry, and inflammatory status is evaluated weekly using C-reactive protein (CRP) and procalcitonin. Daily protein intake is recorded and expressed in grams per kilogram of body weight per day. Comparative analyses will evaluate outcomes according to protein intake achieved during the second week of ICU stay (>1.3 vs. ≤1.3 g/kg/day).

SUMMARY:
Survival of critically ill patients has improved, resulting in a growing population of chronically critically ill (CCI) individuals with prolonged organ dysfunction, mechanical ventilation, and high morbidity. While nutritional guidelines during the acute phase are well established, evidence on protein intake in CCI patients is limited. Inflammation may influence metabolic responses and clinical outcomes, highlighting the need for prospective studies.

The MetaChronic Study is a single-center, prospective cohort designed to describe metabolic trajectories and evaluate the effect of protein intake on outcomes in critically ill adults. Resting energy expenditure will be measured by serial indirect calorimetry, protein and caloric intake will be recorded weekly, and inflammation will be assessed using C-reactive protein (CRP) and procalcitonin. Secondary objectives include subgroup analyses, assessment of protein delivery routes, and exploration of interactions between protein intake, caloric intake, and inflammation.

DETAILED DESCRIPTION:
This single-center, longitudinal observational study enrolls critically ill adults who require invasive mechanical ventilation (IMV) for at least 48 hours and remain in the Intensive Care Unit (ICU) for more than 7 days. Participants are followed in-hospital for up to 42 days after ICU admission, unless discharged, deceased, or unable to continue accurate nutritional monitoring due to transition to oral feeding for nutritional purposes. The final assessment occurs on Day 90 after onset of critical illness, when functional status is evaluated using the Portuguese validated version of the EuroQol 5-Dimension Questionnaire (EQ-5D), administered either by telephone or in person depending on patient location.

Baseline characterization includes:

* Demographic information (age, sex)
* Pre-ICU hospitalization days
* Nutritional risk assessed with the modified Nutrition Risk in the Critically Ill (NUTRIC) score (without interleukin-6)
* Category of critical illness (septic with/without abdominal surgery, trauma with/without head injury, neurocritical, and other categories)
* Severity upon ICU admission measured by the Simplified Acute Physiology Score II (SAPS II)

Metabolic assessment is performed using serial indirect calorimetry beginning on Day 7 of ICU stay and repeated one to three times per week up to Day 42 or until hospital discharge. Feasibility requires absence of air leaks in the respiratory system. For patients on invasive mechanical ventilation (IMV), measurements follow device requirements (fraction of inspired oxygen < 70% and positive end-expiratory pressure < 12 cmH₂O); for spontaneous ventilation, measurements are obtained in canopy mode at FiO₂ 21%. Weekly metabolic values are calculated as the average of available measurements.

Protein intake is recorded according to routine clinical practice and quantified weekly after Day 7, expressed in grams (g) per kilogram of adjusted body weight per day (g/kg/day). Protein delivered as amino acids is converted to grams of protein using a standard factor (100 g hydrolyzed protein = 83 g amino acids). Total caloric intake is also quantified weekly, including enteral and parenteral nutrition as well as non-nutritional caloric sources such as glucose-containing solutions and propofol.

Inflammatory status is assessed weekly using C-reactive protein (CRP) and procalcitonin measurements.

Patients are monitored according to routine clinical practice, and comparative analyses will evaluate outcomes according to protein intake achieved during the second week of ICU stay (>1.3 vs. ≤1.3 g/kg/day). Outcomes include:

* Duration of invasive mechanical ventilation (days)
* Days alive and out of the ICU to Day 90 (days)
* Days alive and out of the hospital to Day 90 (days)
* Need for tracheostomy (Yes/No); if yes, possibility of decannulation (Yes/No)
* Duration of tracheostomy (days)
* Mortality at 28 days, in ICU, in-hospital, and at 90 days
* Number of infections to Day 30 (defined as the number of infectious agents, not deemed colonization, in biological samples obtained per local standard practice)
* Discharge destination (institution/home)
* Functional outcome at Day 90 assessed using the EuroQol 5-Dimension Questionnaire (EQ-5D)

ELIGIBILITY:
Inclusion Criteria:

* Adult critically ill patients admitted to Intensive Care Unit > 7 days
* Invasive mechanical ventilation (IMV) > 48 hours

Exclusion Criteria:

* Active oncological disease
* Neuromuscular diseases
* Confirmed or predicted Glasgow Coma Score < 10 at 14 days in Intensive Care Unit
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include adult critically ill patients admitted to intensive care who meet the eligibility criteria described.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2024-03-15 (Actual); Primary Completion 2024-06-15 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Resting Energy Expenditure (REE) | From Day 7 of Intensive Care Unit stay through Day 42 or until Intensive Care Unit, whichever occurs first.
  Resting energy expenditure will be measured by indirect calorimetry using a calorimeter, which calculates energy expenditure in kilocalories (Kcal) per day from oxygen consumption and carbon dioxide production. Serial measurements will characterize metabolic trajectories during prolonged critical illness.

SECONDARY OUTCOMES:
Mortality | At Intensive Care Unit (ICU) discharge; at Day 28 after ICU admission; at hospital discharge; at Day 90 after ICU admission.
  Mortality at multiple time points. Values: Alive/Dead.
Duration of Invasive Mechanical Ventilation | From endotracheal intubation to extubation or transition to intermittent ventilation via tracheostomy, up to Day 42 of ICU stay.
  Number of days the patient requires invasive mechanical ventilation, from the time of endotracheal intubation until extubation or transition to intermittent ventilation via tracheostomy.
Protein Intake | From Day 7 of Intensive Care Unit stay through Day 42 or until Intensive Care Unit discharge, whichever occurs first
  Daily protein intake will be recorded based on routine clinical practice. Values will be reported in grams per kilogram of body weight per day (g/kg/day). Weekly averages will be calculated to characterize protein provision during prolonged critical illness.
Tracheostomy Duration | From tracheostomy insertion through decannulation, up to 90 days.
  Number of days from tracheostomy insertion to decannulation, if performed.
Number of Infections | From Intensive Care Unit admission through Day 30
  Number of infections diagnosed within 30 days of Intensive Care Unit admission. Defined as the number of infectious agentes, not deemed to be colonization, in biological samples performed in accordance with local standard practice
Days Alive and Out of the Intensive Care Unit | From Intensive Care Unit admission through Day 90.
  Number of days the patient is alive and not in the Intensive Care Unit, calculated from Intensive Care Unit admission through Day 90.
Days Alive and Out of the Hospital | From hospital admission through Day 90.
  Number of days the patient is alive and not in the hospital, calculated from hospital admission through Day 90.
Discharge Destination | At Day 42 after Intensive Care Unit admission
  Discharge destination among survivors. Values: Home/Institution (for example, rehabilitation facility).
Functional Status at 90 Days | At Day 90 after Intensive Care Unit admission
  Patient functional status measured using the EQ-5D scale among survivors at Day 90.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Binnie, Study Chair — Universidade do Algarve
Locations (1):
- Algarve, Faro, Portugal

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) to be shared include: de-identified demographic and clinical variables (age, sex, diagnosis, severity scores), nutritional data (caloric and protein intake, feeding route), indirect calorimetry results, inflammatory markers (C-reactive protein, procalcitonin), and outcome variables (ICU/hospital length of stay, mortality).
Supporting Information: Study Protocol
Time Frame: Beginning 3 months after publication and ending 2 years after the publication of results
Access Criteria: De-identified individual participant data and supporting documents (protocol, analysis plan, CRFs) will be made available as supplementary material to the publication and can also be shared with qualified researchers upon reasonable request. Access requires submission of a research proposal and signing a data use agreement to ensure confidentiality and compliance with ethical regulations.

REFERENCES:
- [Background] Moonen HPFX, Beckers KJH, van Zanten ARH. Energy expenditure and indirect calorimetry in critical illness and convalescence: current evidence and practical considerations. J Intensive Care. 2021 Jan 12;9(1):8. doi: 10.1186/s40560-021-00524-0. PMID 33436084